CLINICAL TRIAL: NCT06349369
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on Inflammatory Biomarkers in Chronic Schizophrenia: A Randomised Double-Blind Controlled Trial.
Brief Title: Effect of tDCS on Inflammatory Biomarkers in Chronic Schizophrenia
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Debadatta Mohapatra, Associate Prof, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG Thesis/2023-24/105
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Chronic Schizophrenia
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): the cathode will be located over a point midway between T3 and P3 (left temporo-parietal junction, assumed to correspond to a region including BA 22, 39, 40, 41, and 42, depending on the patient) and the anode will be placed with the middle of the electrode over a point midway between F3 and FP1 (left prefrontal cortex: dorsolateral prefrontal cortex, assumed to correspond to a region including Brodmann's areas [BA] 8, 9, 10, and 46, depending on the patient).The transcranial brain stimulation will be given 2 sessions per day for 10 days, in which 20 minutes of stimulation with an inter-session interval of 3 hours.
  Interventions: Device: transcranial direct current stimulation
- Sham control group (Sham Comparator): To Maximize the stimulatory effects 1mA current will be applied for the first 30 seconds, to provide the initial sensation of real stimulation and then the current will be stopped, thus minimizing the stimulatory effects.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS is a non-invasive neuromodulation technique that has gained attention for its potential to influence neural activity and address cognitive and functional deficits in individuals with schizophrenia. It involves applying a weak direct electrical current to the scalp, which can increase or decrease the excitability of underlying brain regions.

SUMMARY:
The study is a randomized, double-blind, parallel-arm, sham-controlled trial that aims to compare the effects of transcranial direct current stimulation (tDCS) versus sham stimulation on inflammatory markers (IL-6 and TNF-alpha) and clinical outcomes (PANSS, AHRS, CGI-SCH, GAF) in patients with chronic schizophrenia over 10 days of treatment. The primary objective is to assess changes in IL-6 levels, while secondary objectives include evaluating changes in TNF-alpha, symptom scales, and adverse events. The study will be conducted at the psychiatry department of AIIMS Bhubaneswar, with 60 patients aged 18-60 years with moderate-to-severe schizophrenia symptoms randomized to receive either active tDCS (cathode over left temporo-parietal junction, anode over left dorsolateral prefrontal cortex) or sham stimulation. The researchers hope to elucidate the potential immunomodulatory effects of tDCS and its impact on symptoms in chronic schizophrenia, which may lead to more targeted, multifaceted interventions to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients clinically diagnosed with schizophrenia (F20 according to ICD-11) for a period more than 2 years receiving antipsychotics.

2. Moderate to severe symptoms (PANSS score >75 and/or CGI-SGH score >4) 3. Patients of both sex 18-60 years 4. Right-handed. 5. Legally authorized representative (LAR) giving voluntary written consent for participation in the study.

Exclusion Criteria:

* 1. Patients with chance of pregnancy. 2. Any psychiatric emergency (e.g. suicidal risk, catatonia, prolonged nutritional deprivation) or others (e.g.: aggression or excitement) 3. Co-morbid neurological disease: i) History of migraine. ii) History of seizure/epilepsy. iii) History of head trauma or organic disease.

  4. Any contraindication to tDCS procedure: i) Injury or local lesion in the scalp/head ii) Metallic implants in the head iii) Implanted brain medical devices 5. Left-handed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Change in the IL-6 levels | 10 days

SECONDARY OUTCOMES:
Change in the TNF alpha levels. | 10 days
Change in the Positive and Negative syndrome Scale | 5 days and 10 days
  score 1- absent symptoms Score 7- extreme symptoms
Change in the Auditory hallucination rating scale | 5 days and 10 days
  score 0- No Auditory hallucination Score 9- Severe Auditory hallucination
Change in the Clinical global impression- Schizophrenia scale | 5 days and 10 days
  score 0- not assessed score 7- extremely ill patients
Change in the Global Assessment of Functioning scale | 5 days and 10 days
  score 0- inadequate information score 100- No symptoms
To compare the adverse events reported in both control and intervention groups. | 5 days and 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Result] Vaseghi B, Zoghi M, Jaberzadeh S. A meta-analysis of site-specific effects of cathodal transcranial direct current stimulation on sensory perception and pain. PLoS One. 2015 May 15;10(5):e0123873. doi: 10.1371/journal.pone.0123873. eCollection 2015. PMID 25978673
- [Result] Xu H, Zhou Y, Wang J, Liang Z, Wang Y, Wu W, Liu Y, Liu X, Zhang X, Huo L. Effect of HD-tDCS on white matter integrity and associated cognitive function in chronic schizophrenia: A double-blind, sham-controlled randomized trial. Psychiatry Res. 2023 Jun;324:115183. doi: 10.1016/j.psychres.2023.115183. Epub 2023 Mar 27. PMID 37028258
- [Result] Hafner H, an der Heiden W. Epidemiology of schizophrenia. Can J Psychiatry. 1997 Mar;42(2):139-51. doi: 10.1177/070674379704200204. PMID 9067063
- [Result] Schennach R, Riedel M, Obermeier M, Spellmann I, Musil R, Jager M, Schmauss M, Laux G, Pfeiffer H, Naber D, Schmidt LG, Gaebel W, Klosterkotter J, Heuser I, Maier W, Lemke MR, Ruther E, Klingberg S, Gastpar M, Moller HJ. What are residual symptoms in schizophrenia spectrum disorder? Clinical description and 1-year persistence within a naturalistic trial. Eur Arch Psychiatry Clin Neurosci. 2015 Mar;265(2):107-16. doi: 10.1007/s00406-014-0528-2. Epub 2014 Sep 27. PMID 25261210
- [Result] Palm U, Keeser D, Hasan A, Kupka MJ, Blautzik J, Sarubin N, Kaymakanova F, Unger I, Falkai P, Meindl T, Ertl-Wagner B, Padberg F. Prefrontal Transcranial Direct Current Stimulation for Treatment of Schizophrenia With Predominant Negative Symptoms: A Double-Blind, Sham-Controlled Proof-of-Concept Study. Schizophr Bull. 2016 Sep;42(5):1253-61. doi: 10.1093/schbul/sbw041. Epub 2016 Apr 20. PMID 27098066
- [Result] Siskind D, Siskind V, Kisely S. Clozapine Response Rates among People with Treatment-Resistant Schizophrenia: Data from a Systematic Review and Meta-Analysis. Can J Psychiatry. 2017 Nov;62(11):772-777. doi: 10.1177/0706743717718167. Epub 2017 Jun 28. PMID 28655284
- [Result] Muller N, Weidinger E, Leitner B, Schwarz MJ. The role of inflammation in schizophrenia. Front Neurosci. 2015 Oct 21;9:372. doi: 10.3389/fnins.2015.00372. eCollection 2015. PMID 26539073
- [Result] Huarcaya-Victoria J, Villarreal-Rao B, Luna M, Rojas-Mendoza W, Alarcon-Ruiz CA, Villarreal-Zegarra D, Vilela-Estrada AL, Ramirez S. Factors Associated with Mental Health Outcomes in Hospital Workers during the COVID-19 Pandemic: A Mixed-Methods Study. Int J Environ Res Public Health. 2022 Apr 28;19(9):5346. doi: 10.3390/ijerph19095346. PMID 35564741
- [Result] Thair H, Holloway AL, Newport R, Smith AD. Transcranial Direct Current Stimulation (tDCS): A Beginner's Guide for Design and Implementation. Front Neurosci. 2017 Nov 22;11:641. doi: 10.3389/fnins.2017.00641. eCollection 2017. PMID 29213226
- [Result] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Result] Valiengo LDCL, Goerigk S, Gordon PC, Padberg F, Serpa MH, Koebe S, Santos LAD, Lovera RAM, Carvalho JB, van de Bilt M, Lacerda ALT, Elkis H, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation for Treating Negative Symptoms in Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):121-129. doi: 10.1001/jamapsychiatry.2019.3199. PMID 31617873
- [Result] Goerigk S, Cretaz E, Sampaio-Junior B, Vieira ELM, Gattaz W, Klein I, Lafer B, Teixeira AL, Carvalho AF, Lotufo PA, Bensenor IM, Buhner M, Padberg F, Brunoni AR. Effects of tDCS on neuroplasticity and inflammatory biomarkers in bipolar depression: Results from a sham-controlled study. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Mar 8;105:110119. doi: 10.1016/j.pnpbp.2020.110119. Epub 2020 Oct 4. PMID 33022345
- [Result] Agarwal SM, Shivakumar V, Bose A, Subramaniam A, Nawani H, Chhabra H, Kalmady SV, Narayanaswamy JC, Venkatasubramanian G. Transcranial direct current stimulation in schizophrenia. Clin Psychopharmacol Neurosci. 2013 Dec;11(3):118-25. doi: 10.9758/cpn.2013.11.3.118. Epub 2013 Dec 24. PMID 24465247